CLINICAL TRIAL: NCT04424459
Title: Evaluation of an Opioid Decrease Strategy in Chronic Pain Patients at the Pain Assessment and Treatment Center in Montpellier: Prospective Study Over 6 Months.
Brief Title: Evaluation of an Opioid Decrease Strategy in Chronic
Acronym: EODSCPP
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0132
Record Dates: First submitted 2020-05-28; First posted 2020-06-11 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Chronic Pain
Keywords: Opioid analgesics; Opioid use disorders; Prescription drug abuse; treatments Prevention Identification
MeSH Terms: conditions — Chronic Pain; Opioid-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — NC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients included from 10/01/19 to 12/31/19.: Patients included from 10/01/19 to 12/31/19. (the study will be extended to a larger number of patients according to the first results), continued according to the first results. DCNC patients treated at the Montpellier Pain Assessment and Treatment Center hospitalized during the period from 10/01/19 to 12/31/19, for misuse of opioid treatment.
  Interventions: Drug: opioid withdrawal

INTERVENTIONS:
Drug: opioid withdrawal — The data retrieved from the patient will be encrypted and there will also be written data or written in binary form. They will be used to create an Excel table which allows me to list the data on D1 then on M + 3 then on M + 6 in order to evaluate the evolution of these data over a time interval of 6 months and this is which will be used as support in my thesis in pharmacy.

SUMMARY:
Increase in the consumption of analgesics observed in many countries with a mediatic crisis resulting in an increasingly frequent wish of patients to wean themselves from opiates. A recent update (B. Rolland 2017) suggests that upon initiation of an opioid analgesic treatment, the patient should be informed of the risk of opioid dependence and misuse. There is no clearly validated decay scheme in the event of dependence in patients with Chronic Non-Cancer Pain.

Hypotheses:

* Possibility of a rapid decrease in opioid analgesic treatments at DCNC sensitized to the risk of DOP and MOP. (Protocol implemented: Multidisciplinary assessment, workshops and information sheet on chronic pain, treatments and risk of DOP, pharmacological and nonpharmacological adaptation)
* Highlight the need for additional information from patients and prescribers on the risk of DOP and MOP in DCNC.

DETAILED DESCRIPTION:
Main objective: Check if the rapid to semi-rapid regimen (- 25 to -60% dosage in 5 days of HDS) of opioid analgesics, without the use of methadone or buprenorphine agonists, in the case of DCNC at the CETD in Montpellier is efficient in the medium term (6 months).

Secondary objective:

* With our inclusion questionnaire we wanted to check if the patients had been made aware of the risk of opiate dependence and misuse.
* Detect the conditions of prescriptions that can promote the misuse of opiates.
* Evaluating the different components of residual pain at 6 months (type, intensity, anxiety component and depression, function).

ELIGIBILITY:
Inclusion criteria:

* chronic pain patient
* major
* supported at CETD

Exclusion criteria:

-patient with physical and mental incapacity to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: DCNC patients treated at the Montpellier Pain Assessment and Treatment Center hospitalized during the period from 10/01/19 to 12/31/19, for misuse of opioid treatment.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Change of the dosage of opioid and co-analgesic treatments | 3 months and 6 months
  Change of the dosage of opioid and co-analgesic treatments

SECONDARY OUTCOMES:
Measuring quality of life | Inclusion, 3 and 6 months
  interview with the patient

CONTACTS AND LOCATIONS:
Overall Officials: Théa GENDARME, MD, PharmD, MSc, Principal Investigator — UH Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC